CLINICAL TRIAL: NCT05009017
Title: The Safety Study of Bevacizumab Biosimilars in the Real World
Brief Title: Multi-Centre, Observational Study on Safety of Bevacizumab Biosimilars in Clinical Practice Among Chinese Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Guohui Li, Pharmacy, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC2863
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Biosimilar
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Biosimilar group
  Interventions: Drug: Bevacizumab
- Originator group
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Patients with colorectal cancer or lung cancer who use originator or biosimilar of bevacizumab

SUMMARY:
Monoclonal antibody drugs are expensive, and the listing of biosimilar drugs can help increase the availability and lower prices of biologic drugs, and can better meet the public's demand for biotherapeutic products. The first bevacizumab biosimilar in China was launched in December 2019. Although monoclonal antibody biosimilar drugs are similar to the original drug in terms of quality, safety and effectiveness, their production process may be different from the original drug, and their clinical application cannot be completely equivalent to the original drug. Especially after the market is applied to a wider patient population, the safety and effectiveness are more worthy of attention. This study started from the perspective of pharmacy. Three hospitals in China participated in the real-world safety assessment of bevacizumab biosimilars. An observational cohort study design was adopted to include all cases of lung cancer and colorectal cancer using bevacizumab biosimilars and original drugs during the study period, and the propensity score matching was used to reduce the influence of confounding factors and conduct safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* ①Inpatients diagnosed with non-small cell lung cancer or colorectal cancer; ②Bevacizumab biosimilars or original drugs were used for treatment during the study period.

Exclusion Criteria:

* ①Age<18 years old; ②Person who has used bevacizumab within six months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients in 3 study hospitals diagnosed with non-small cell lung cancer or colorectal cancer using originator or biosimilar of bevacizumab
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse drug reactions | 12 months
  Severity of adverse drug reactions

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Wenzhou Zhang, Zhengzhou, Henan